CLINICAL TRIAL: NCT06342050
Title: Socioecological Factors Associated With Ethnic Disparities in Bariatric Surgery Utilization and Post-Operative Weight Loss (Substudy)
Brief Title: Socioecological Factors Associated With Ethnic Disparities in Bariatric Surgery Utilization and Post-WLS
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Benjamin Schneider, Associate Professor & Division Chief - Bariatric & Foregut Surgery, University of Texas Southwestern Medical Center
Other Study IDs: STU-2023-0548; R01MD011686 (NIH)
Record Dates: First submitted 2024-02-22; First posted 2024-04-02 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: Weight loss surgery; Bariatric surgery; Gut Microbiome; Blood Microbiome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 2 blood sample tubes collected at the same timepoint and 1 stool sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WLS non-completers: Participants who did not have WLS as part of the main study
- WLS completers: Participants who had WLS as part of the main study

SUMMARY:
The goal of this cross-sectional observational study is to examine potential relationships between the blood and gut microbiota of patients with obesity before and after weight loss surgery (WLS) and evaluate potential ethnic differences in the blood and gut microbiotas before and after the WLS.

The main aims / objectives of this sub-study are:

* Aim 1. Compare the relationship between the blood and the gut microbiomes among a sample of (1) pre-WLS and (2) 6-month post-WLS participants.

Hypothesis: Blood bacterial composition will resemble that of the gut microbiome among pre-WLS participants. Because the effect of WLS on the blood microbiome is not known, our post-WLS results will be mostly exploratory.

* Aim 2. Determine racial differences in the blood microbiome of the pre- and post-WLS groups.

Hypothesis2: Ethnic differences will be detected in both the pre- and post-WLS groups.

DETAILED DESCRIPTION:
A subgroup of participants from the main study will be invited to participate in a cross-sectional sub study evaluating the relationship between blood and gut microbiotas. A total of 100 participants will be recruited, 50 participants will be recruited from the "non-completers" and the other 50 participants will be recruited from the "6 months post-WLS" follow-up group of our main project.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* Will belong to either Non-Hispanic Whites (NHW) or Non-Hispanic Blacks (NHB) ethnic groups
* "No-WLS" participants will have a BMI >35 kg/m2 (threshold BMI for WLS) whereas "6 months post-WLS" participants will have no BMI requirements.

Exclusion Criteria:

* Having taken antibiotics in the previous 6 months;
* Metformin, proton pump inhibitors, probiotics, or prebiotics in the previous month;
* Currently following a vegetarian diet;
* Pregnancy;
* Having any infection in the previous month; and
* Having a comorbid disease that might alter the blood microbiome composition (e.g., renal failure) or the intestinal permeability (e.g., IBS).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Investigators will recruit in the following manner:
  * Non-surgery participants from the "non-completers" group from the main study
  * Participants who had bariatric surgery 6 months prior to their enrollment into this sub study, will be recruited from the "early and late completers" in the main study. If additional participants are needed, particularly due to strict ethnic requirements (limited to NHW and NHB), first, invitation emails will be sent to the Weight Wellness Clinic patients, and if recruiting at the expected rate continues to be an issue, advertisements through IRB-approved flyers on social media or in the clinic setting will be posted.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Gut Microbial Composition | Stool samples will be collected at one time point only, within a week to their in person appointment.
  Gut microbial composition will be measured by performing whole metagenome sequencing in samples previously stored in Zymo stool collection tubes.
Blood Microbial Composition | Blood samples will be collected in fasting conditions at the Baseline visit.
  Blood microbial composition will be measured by performing 16S rRNA (ribosomal ribonucleic acid) in blood samples previously stored in Zymo blood collection tubes.
Body Weight (kg) | Baseline
  Body weight will be measured with a calibrated SECA scale.
Body Height (meters) | Baseline
  Body height will be measured with a stadiometer.
Fat Mass (Kg) | Baseline
  Body fat mass will be measured by using the SECA mBCA 515.
Fat-free Mass (Kg) | Baseline
  Fat-free mass will be measured by using the SECA mBCA 515.
Body water (%) | Baseline
  Body water percentage will be measured by using the SECA mBCA 515.
Skeletal Muscle Mass (kg) | Baseline
  Skeletal muscle mass will be measured by using the SECA mBCA 515.
Fasting Glucose (mg/dL) | Baseline
  Fasting glucose will be measured after a 12h fast.
Fasting Insulin (mIU/L) | Baseline
  Fasting insulin will be measured after a 12h fast.
Lipopolysaccharides (%) | Baseline
  Lipopolysaccharides will be measured after a 12h fast.
Lipopolysaccharides binding protein (mIU/L) | Baseline
  Lipopolysaccharides binding protein will be measured after a 12h fast.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Schneider, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT06342050/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT06342050/ICF_001.pdf